CLINICAL TRIAL: NCT05089994
Title: Comparison of Two Approaches of Quadratus Lumborum Block for Post-operative Analgesia in Radical Cystectomy: Prospective-randomized Clinical Trial
Brief Title: Comparison of Two Approaches of Quadratus Lumborum Block for Post-operative Analgesia in Radical Cystectomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hassan mostafa abdelbaky ahmed, Comparison of Two Approaches of Quadratus Lumborum Block for Post-operative Analgesia in Radical Cystectomy, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 01060264751
Record Dates: First submitted 2021-05-22; First posted 2021-10-22 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-06

CONDITIONS: Quadratus Lumborum Block

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (QLBA) will include 30 patients (Experimental): will receive ultrasound-guided anterior approach quadratus lumborum block
  Interventions: Procedure: US guided injection
- Group 2 (QLBI)will include 30 patients. (Experimental): received ultrasound-guided intramuscular quadratus lumborum.
  Interventions: Procedure: US guided injection

INTERVENTIONS:
Procedure: US guided injection — using 2.5mg/kg of 0.25% bupivacaine diluted in a 20 mL syringe of normal saline , received ultrasound-guided quadratus lumborum.

SUMMARY:
To compare the postoperative analgesic effect of two ultrasound guided approaches of quadratus lumborum block (QLB) (anterior and intramuscular) for radical cystectomy.

DETAILED DESCRIPTION:
The quadratus lumborum block (QLB) is one of the abdominal wall block techniques used to anesthetize thoracolumbar nerves . The QLB technique was described initially by Blanco et al. in 2007 (not published), then reported initially by Kadam in 2013. Since then, QLB has evolved with the development of the ultrasound-guided nerve block. To date, several randomized controlled trials have reported effective postoperative analgesia, with non-intramuscular QLB for cesarean sections, laparoscopic gynecologic surgery and hip hemiarthroplasty .

The intramuscular QLB (QLBi) technique was first reported by. This approach is different from others in tubouchi for QLB; although the injection target sites of the other approaches are planes around the quadratus lumborum muscle, the intramuscular approach penetrates the fascia of the quadratus lumborum muscle, where local anesthetics are injected. Therefore, QLBi is relatively easier to perform compared with other QLB approaches.

The incidence of urinary bladder cancer in the Middle East and Africa is greater in areas with high rather than low SH prevalence.

ELIGIBILITY:
Inclusion Criteria:

* Age: 40-70years.

  * BMI: 20-30 kg.m2
  * Sex: both males and females.
  * American Society of Anesthesiologists (ASA )physical status: I-III.
  * Operation: radical cystectomy

Exclusion Criteria:

* • Patient's refusal to participate in the study.

  * known allergy to local anesthesia (LA),
  * coagulopathy or thrombocytopenia,
  * body mass index (BMI) above 30 kg .m 2, and infection at site of injection.
  * Chronic pain syndromes,
  * Prolonged opioid medication,
  * Patients on regular use of analgesic or who received analgesic 24 h before surgery

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-10-06 (Actual); Primary Completion 2024-09-04 (Estimated); Study Completion 2024-09-25 (Estimated)

PRIMARY OUTCOMES:
Evaluate the first call for rescue analgesia | 24hours after recovery From anesthesia
  The time of the first call of analgesia is recorded

SECONDARY OUTCOMES:
Total doses of morphine required | 24hours after recovery from anesthesia
  Doses of morphine required postoperative

CONTACTS AND LOCATIONS:
Locations (1):
- Assuit university urology hospital, Asyut, Egypt